CLINICAL TRIAL: NCT01381029
Title: A Study to Examine Immunological Response in HIV-Infected Patients Receiving the Seasonal Influenza Vaccine
Brief Title: Immune Response to Seasonal Influenza Vaccine in HIV Infected Individuals
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB080911
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Influenza, Human; Human Immunodeficiency Virus I Infection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV positive: HIV positive, receiving Influenza vaccine as standard of care.

SUMMARY:
Investigators in the Division of Infectious Diseases are carrying out a study to determine if human immunodeficiency virus (HIV)-seropositive patients receiving the Seasonal Influenza vaccination develop an adequate antibody response. The study group will consist of individuals seen in the Infectious Diseases Clinic who are HIV-seropositive and receive the Seasonal Influenza vaccine.

DETAILED DESCRIPTION:
This is a study to establish the immunologic response in HIV-seropositive individuals to the FDA approved seasonal influenza vaccine when it is available. HIV-seropositive individuals seen in the Infectious Diseases Clinic at George Washington University, Medical Faculty Associates and receive this vaccination, on label, as part of standard of care will be invited to participate.

The study will require a 10-ml sample of whole blood to be drawn from each participant prior to the dose of the seasonal influenza vaccine and at 3 weeks after the vaccine dose and at 3 months after the vaccine dose. No additional samples are envisioned. Serum will be separated and will frozen and stored in the Clinical Trials Unit until all patient samples have been obtained. At that time the antibody levels to the vaccine antigens will be measured.

Data that will be collected from the subject's medical record includes the following:

* Age, gender, race
* CD4 count
* HIV viral load
* History of prior influenza immunization including the 2009-2010 trivalent vaccine
* HIV antiviral medication history

Data that will be collected from the subject during participation in study

* Antibody levels prior to vaccination
* Dose date of the seasonal influenza vaccination
* Antibody levels 3 weeks after the vaccination

ELIGIBILITY:
Inclusion Criteria:

* Males or female patients ages 18 or older
* Diagnosis of HIV infection
* No contraindications to being able to receive influenza vaccine by the treating physician
* No acute active illness
* Able to provide informed consent

Exclusion Criteria:

* Previous history of hypersensitivity reaction to influenza vaccine
* Unable to return for follow-up blood draw

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive individuals receiving influenza vaccine as part of standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2009-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in antibody levels | Pre-, 3 weeks post-, 3 months post- vaccine
  The primary endpoint will be to measure the change from baseline in vaccine-strain specific antibody levels. Titers of > or = 40 U will be considered protective and a > 4-fold rise in antibody titer will be considered an adequate response in previously antibody-negative patients. Data from this study will assist in defining the efficacy of the influenza vaccine in the HIV-infected population and the ability of HIV-infected patients to generate an appropriate immune response, as well as maintain an appropriate response, to the influenza vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Siegel, MD, Principal Investigator — George Washington University
Locations (1):
- Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No